CLINICAL TRIAL: NCT01966107
Title: Double-blind, Randomized, Placebo-controlled, Parallel-group, Phase IV Study to Evaluate the Effect of Aclidinium Bromide on Long-term Cardiovascular Safety and COPD Exacerbations in Patients With Moderate to Very Severe COPD (ASCENT COPD)
Brief Title: Evaluate the Effect of Aclidinium Bromide on Long-term Cardiovascular Safety and Exacerbations in Moderate to Very Severe COPD Patients.
Acronym: ASCENT COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6560C00002; LAS-MD-45 (Other: Forest Research)
Record Dates: First submitted 2013-10-16; First posted 2013-10-21 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease; Moderate to Very Severe COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aclidinium Bromide (Experimental): Two-week washout/run-in period [for patients on a long-acting muscarinic antagonist (LAMA)] followed by a maximum of 36-month double-blind treatment period.
  Interventions: Drug: Aclidinium Bromide
- Placebo (Placebo Comparator): Two-week washout/run-in period [for patients on a long-acting muscarinic antagonist (LAMA)] followed by a maximum of 36-month double-blind treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium Bromide — 400 μg, twice per day, oral administration via a multi-dose dry-powder inhaler (DPI)
  Arms: Aclidinium Bromide
Drug: Placebo — Dose matched placebo, twice per day, oral administration via a multi-dose dry-powder inhaler (DPI)
  Arms: Placebo

SUMMARY:
The Objectives of this study are to assess the safety of Aclidinium bromide on major adverse cardiovascular events (MACE), to assess the overall safety of Aclidinium bromide and to assess whether Aclidinium bromide reduces moderate or severe COPD exacerbations. This study is a double-blind, randomized, placebo controlled, parallel-group study to evaluate the effect of Aclidinium bromide on the cardiovascular safety and COPD exacerbations in patients with moderate to very severe COPD, as defined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female outpatients ≥ 40 years of age
* 2. Current or former cigarette smokers with a smoking history of at least 10 pack-years
* 3. A diagnosis of stable, moderate to very severe COPD (GOLD, 2015) with a post-bronchodilator FEV < 80% FEV1/forced vital capacity (FVC) ratio < 70%
* 4. Must have at least one of the following 4 criteria:

  1. Documented cerebrovascular disease (stroke or transient ischemic attack, carotid stenosis)
  2. Documented coronary artery disease (angina, MI, angioplasty/stent/bypass)
  3. Documented peripheral vascular disease or history of claudication
  4. At least 2 of the following atherothrombotic risk factors as determined by the PI:

     1. Male ≥ 65 years or female ≥ 70 years
     2. Diabetes
     3. Dyslipidemia
     4. Hypertension
     5. Waist circumference inches males ≥ 40 in or in females ≥ 38 inches
     6. Evidence of renal dysfunction (eGFR < 60) and microalbuminuria (eGFR is based on modification of diet in renal disease [MDRD] equation, microalbuminuria is defined as ≥ 30-300 mcg/mg creatinine on a spot urine or ≥30 mg creatinine on a 24hr urine test)
* 5. Maintained stable respiratory medications for 2 weeks prior to randomization (Appendix II)
* 6. Able to perform pulmonary function test (PFT) maneuvers and follow study procedures
* 7. Women of childbearing potential must have a negative serum β-human chorionic gonadotropin (HCG) pregnancy test at Visit 1A and be practicing medically acceptable method of contraception. Otherwise, female patients should be at least 1 year postmenopausal, surgically sterile (defined as having a hysterectomy or tubal ligation).
* 8. Should understand study procedures and be willing to participate in the study as indicated by signing the ICF

Exclusion Criteria:

* 1. Significant diseases other than COPD or cardiovascular disease (e.g., metastatic cancer) which, in the opinion of the PI, may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* 2. Unstable or life threatening cardiovascular disease or COPD as determined by the PI
* 3. Patients with comorbid lung disease such as asthma, cystic fibrosis, bronchiectasis, interstitial lung disease, or pulmonary thromboembolic disease
* 4. Planned lung transplant or lung volume reduction surgery
* 5. Currently treated with a combination of LAMA and LABA/ICS therapy.
* 6. Malignancy for which patient has undergone resection, radiation therapy or chemotherapy within 5 years prior to screening. Patients with treated basal cell and squamous cell (skin) carcinoma are allowed
* 7. Respiratory infection or COPD exacerbation at Screening and/or within 4 weeks prior to screening
* 8. Uncontrolled infection resulting from human immunodeficiency virus (HIV) and/or active hepatitis
* 9. Reported history of drug or alcohol abuse within the past 12 months
* 10. History of hypersensitivity reaction to inhaled anticholinergics, sympathomimetic amines, or inhaled medication or any component thereof (including report of paradoxical bronchospasm)
* 11. History of acute urinary retention, treatment refractory benign prostatic hyperplasia (BPH), bladder neck obstruction, or narrow-angle glaucoma (Note: Patients with controlled, stable BPH are not excluded)
* 12. Patients unable to use a multidose DPI or a pressurized metered-dose inhaler
* 13. Treatment with any other investigational drug within 30 days (or 6 half-lives, whichever is longer) before Visit 1A
* 14. Women who are pregnant or breastfeeding
* 15. Use of any prohibited medication listed in Appendix II
* 16. Employee or immediate relative of an employee of AstraZeneca, any of its affiliates or partners, or the study center

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3635 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R. Chapman, MD MSc FRCPC FACP FCCP, Principal Investigator — GSK-CIHR Research Chair in Respiratory Health Care Delivery,; Robert Wise, MD, Principal Investigator — Johns Hopkins Bayview Medical Center, Asthma and Allergy Center
Locations (364):
- United States (337):
  - Research Site, Birmingham, Alabama
  - Research Site, Florence, Alabama
  - Research Site, Foley, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Encinitas, California
  - Research Site, Escondido, California
  - Research Site, Fresno, California
  - Research Site, Gold River, California
  - Research Site, Huntington Beach, California
  - Research Site, La Mirada, California
  - Research Site, Laguna Hills, California
  - Research Site, Lincoln, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, North Hollywood, California
  - Research Site, Northridge, California
  - Research Site, Palm Desert, California
  - Research Site, Palm Springs, California
  - Research Site, Paramount, California
  - Research Site, Pismo Beach, California
  - Research Site, Port Hueneme, California
  - Research Site, Poway, California
  - Research Site, Rialto, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, San Jose, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Monica, California
  - Research Site, Sherman Oaks, California
  - Research Site, Vista, California
  - Research Site, Westminster, California
  - Research Site, Wildomar, California
  - Research Site, Boulder, Colorado
  - Research Site, Centennial, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Golden, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Bristol, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Wilmington, Delaware
  - Research Site, Bay Pines, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, DeBary, Florida
  - Research Site, DeLand, Florida
  - Research Site, Doral, Florida
  - Research Site, Eustis, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Loxahatchee Groves, Florida
  - Research Site, Maitland, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Naples, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Oviedo, Florida
  - Research Site, Palmetto Bay, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Pinellas Park, Florida
  - Research Site, Plantation, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Santa Rosa Beach, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Sebring, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Duluth, Georgia
  - Research Site, Johns Creek, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Norcross, Georgia
  - Research Site, Oakwood, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Snellville, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Hayden Lake, Idaho
  - Research Site, Idaho Falls, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Gillespie, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, Morton, Illinois
  - Research Site, Normal, Illinois
  - Research Site, North Chicago, Illinois
  - Research Site, O'Fallon, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Elwood, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Council Bluffs, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Lenexa, Kansas
  - Research Site, Pratt, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Bowling Green, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Madisonville, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Crowley, Louisiana
  - Research Site, Eunice, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, Marshall, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Opelousas, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Zachary, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Biddeford, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Elkridge, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Fall River, Massachusetts
  - Research Site, Methuen, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Bingham Farms, Michigan
  - Research Site, Buckley, Michigan
  - Research Site, Caro, Michigan
  - Research Site, Chesterfield, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Rochester, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Stevensville, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, Chesterfield, Missouri
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Fremont, Nebraska
  - Research Site, Grand Island, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Sparks, Nevada
  - Research Site, Belvidere, New Jersey
  - Research Site, Bridgewater, New Jersey
  - Research Site, East Brunswick, New Jersey
  - Research Site, Elizabeth, New Jersey
  - Research Site, Haddon Heights, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Hopewell Jct, New York
  - Research Site, Jamaica, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Wappingers Falls, New York
  - Research Site, Westfield, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Calabash, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Lenoir, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Shelby, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Tabor City, North Carolina
  - Research Site, Whiteville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Delaware, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Yukon, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Beaver, Pennsylvania
  - Research Site, Belle Vernon, Pennsylvania
  - Research Site, Bensalem, Pennsylvania
  - Research Site, Carnegie, Pennsylvania
  - Research Site, Clairton, Pennsylvania
  - Research Site, Downingtown, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Feasterville-Trevose, Pennsylvania
  - Research Site, Jefferson Hills, Pennsylvania
  - Research Site, Levittown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, Uniontown, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Yardley, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Easley, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Hodges, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Pelzer, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Athens, Tennessee
  - Research Site, Chattanooga, Tennessee
  - Research Site, Fayetteville, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Hendersonville, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Smyrna, Tennessee
  - Research Site, Spring Hill, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Boerne, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Corsicana, Texas
  - Research Site, Cypress, Texas
  - Research Site, Dallas, Texas
  - Research Site, Dickinson, Texas
  - Research Site, Duncanville, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Georgetown, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Richardson, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Spring, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Tomball, Texas
  - Research Site, Tyler, Texas
  - Research Site, Waco, Texas
  - Research Site, Webster, Texas
  - Research Site, Midvale, Utah
  - Research Site, Murray, Utah
  - Research Site, Ogden, Utah
  - Research Site, Riverton, Utah
  - Research Site, South Burlington, Vermont
  - Research Site, Abingdon, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Bellingham, Washington
  - Research Site, Everett, Washington
  - Research Site, Port Orchard, Washington
  - Research Site, Spokane, Washington
  - Research Site, Spokane Valley, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Lewisburg, West Virginia
  - Research Site, Morgantown, West Virginia
- Canada (27):
  - Research Site, Edmonton, Alberta
  - Research Site, Kamloops, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, Langley, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, West Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Bridgewater, Nova Scotia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Cornwall, Ontario
  - Research Site, Dorchester, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Thorold, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Chapman KR, Wise RA, Scirica BM, Bhatt DL, Daoud SZ, Lythgoe D, Gil EG. Long-acting antimuscarinic therapy in patients with chronic obstructive pulmonary disease receiving beta-blockers. Respir Res. 2021 Oct 22;22(1):272. doi: 10.1186/s12931-021-01861-2. PMID 34686204
- [Derived] Wise RA, Scirica BM, Bhatt DL, Daoud SZ, Chuecos F, Garcia Gil E, Chapman KR. Efficacy of Aclidinium Bromide According to Baseline Therapy: Post-Hoc Analysis of ASCENT-COPD Randomized Trial. Adv Ther. 2021 Oct;38(10):5381-5397. doi: 10.1007/s12325-021-01878-5. Epub 2021 Sep 15. PMID 34528220
- [Derived] Wise RA, Chapman KR, Scirica BM, Daoud SZ, Lythgoe D, Garcia-Gil E. The Impact of Exacerbation History on the Safety and Efficacy of Aclidinium in Patients with Chronic Obstructive Pulmonary Disease and Increased Cardiovascular Risk: ASCENT-COPD Trial. Int J Chron Obstruct Pulmon Dis. 2021 Mar 18;16:689-699. doi: 10.2147/COPD.S285068. eCollection 2021. PMID 33776428
- [Derived] Wise RA, Chapman KR, Scirica BM, Bhatt DL, Daoud SZ, Zetterstrand S, Reisner C, Gil EG. Effect of Aclidinium Bromide on Major Cardiovascular Events and Exacerbations in High-Risk Patients With Chronic Obstructive Pulmonary Disease: The ASCENT-COPD Randomized Clinical Trial. JAMA. 2019 May 7;321(17):1693-1701. doi: 10.1001/jama.2019.4973. PMID 31063575
- See also: Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4001&filename=AZ-D6560C00002-PXL226451-CSP-amendment5-redacted-Final-31Aug2018_PDFA.pdf
- See also: Statistical Analysis Plan (SAP) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4001&filename=AZ-D6560C00002-PXL226451-SAP-redacted-Final-31Aug2018_PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 522 study centers in North America; 35 centers in Canada and 487 centers in the US. A total of 4000 subjects were planned to be enrolled. A total of 3630 subjects were randomized (1:1) to aclidinium bromide 400 μg twice a day (BID) or placebo BID. Rescue medication (albuterol/salbutamol) was provided for all subjects.
Pre-assignment Details: Informed consent form was signed; inclusion/exclusion, smoking status, electrocardiogram, pregnancy test, Pulmonary function testing, Chronic obstructive pulmonary disease (COPD) exacerbation were assessed. Out of 3635 subjects, 5 subjects were duplicated, who, in violation of protocol entrance criteria, entered the study more than once.
Groups:
- Aclidinium Bromide: Randomized subjects were administered Aclidinium bromide 400 μg BID, once in the morning and once in the evening (approximately 12 hours apart), via a multi-dose dry powder inhalation device (DPI). Subjects on a LAMA (long-acting muscarinic antagonist i.e., inhaled anticholinergics) had to washout 2 weeks prior to randomization.
- Placebo: Randomized subjects were administered placebo, once in the morning and once in the evening (approximately 12 hours apart), via a multi-dose DPI. Subjects on a LAMA (ie, inhaled anticholinergics) had to washout 2 weeks prior to randomization.
Period: Overall Study
Arm/Group | Aclidinium Bromide | Placebo
Started | 1812 | 1818
Full Analysis Set (Subjects included in full analysis set (FAS)) | 1791 | 1798
Completed (Subjects who remained on treatment through this time point) | 1010 | 937
Not Completed | 802 | 881
Not completed — excluded from FAS | 21 | 20
Not completed — discontinued treatment | 345 | 372
Not completed — due to study closure | 164 | 186
Not completed — withdrew from the study | 272 | 303

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) population consisted of all subjects in the Randomized Population who took at least one dose of the double-blind IP (aclidinium bromide or placebo). Subjects were analyzed according to their randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium Bromide | Placebo | Total
Number analyzed (Participants) | 1791 | 1798 | 3589
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (8.5) | 67.2 (8.3) | 67.2 (8.4)
Age, Customized [Count of Participants; unit: Participants]
  >=40 - <60 years | 340 | 325 | 665
  >=60 - <70 years | 724 | 725 | 1449
  >=70 years | 727 | 748 | 1475
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 732 | 752 | 1484
  Male | 1059 | 1046 | 2105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 165 | 138 | 303
  White | 1603 | 1650 | 3253
  Other | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Per Subject Per Year During the First Year of Treatment
Description: The rate (number of events per subject per year) of moderate or severe COPD exacerbations during the first year of treatment based on on-treatment analysis with treatment group, baseline inhaled corticosteroids (ICS) use, baseline COPD severity, history of at least 1 exacerbation in the past year, and smoking status as factors and the log of the exposure time adjusted for the time the subjects experienced exacerbations as an offset variable.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Events per subject per year
Arm/Group | Aclidinium Bromide | Placebo
Number analyzed (Participants) | 1791 | 1798
Events per subject per year | 0.44 [0.40 to 0.50] | 0.57 [0.52 to 0.64]

2. Secondary Outcome: Rate of Hospitalizations Due to COPD Exacerbation Per Subject Per Year During the First Year of Treatment- on Treatment Analysis
Description: To assess whether aclidinium bromide reduces moderate or severe COPD exacerbations. The rate of hospitalization (number of events per subject per year) due to COPD exacerbations during the first year of treatment based on on-treatment analysis with treatment group, baseline ICS use, baseline COPD severity, history of at least 1 exacerbation in the past year, and smoking status as factors and the log of the exposure time adjusted for the time the subjects experienced exacerbations as an offset variable.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Events per subject per year
Arm/Group | Aclidinium Bromide | Placebo
Number analyzed (Participants) | 1791 | 1798
Events per subject per year | 0.07 [0.05 to 0.08] | 0.10 [0.08 to 0.13]
Statistical Analysis 1: Comparison: Aclidinium Bromide vs Placebo; Test type: Superiority; p = 0.006, Negative Binomial Regression model; Rate ratio = 0.65, 95% CI 2-sided [0.48 to 0.89]; A rate ratio <1 represents a favorable outcome for aclidinium bromide 400 μg

3. Secondary Outcome: Number of Participants With Major Adverse Cardiovascular Event (MACE) or Other Serious Cardiovascular Events of Interest - On-study Analysis
Description: To assess the CV safety of aclidinium bromide on MACEs. The number of subjects with an adjudicated MACE or other serious CV events of interest with treatment group, baseline CV severity, and smoking status as factors.
  Other serious CV events included events from Cardiac tachyarrhythmias plus preferred terms (PTs) Tachycardia, Heart rate increase, and Palpitation; Cardiac failure; Bradycardia and PTs Sinus arrest and Sinus bradycardia; Conduction defects; Conditions associated with Central nervous system haemorrhages and cerebrovascular accidents; and selected PTs included in the Other ischemic heart disease.
Time Frame: At Screening, Treatment period (upto 36 months) and Post-treatment follow-up (PTFU)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Aclidinium Bromide | Placebo
Number analyzed (Participants) | 1791 | 1798
Participants
  Number of subjects with events | 168 | 160

4. Primary Outcome: Number of Participants With Major Adverse Cardiovascular Event (MACE) - on Study Analysis
Description: To assess the cardiovascular (CV) safety of aclidinium bromide on MACEs. The number of subjects with an adjudicated composite MACE with treatment group, baseline CV severity, and smoking status as factors. MACE for the analyses was defined as any adjudicated event which was a composite of the total of CV death, non-fatal myocardial infarction (MI), or non-fatal stroke (on-study analysis).
Time Frame: At Screening, Treatment period (upto 36 months) and Post-treatment follow-up (PTFU)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Aclidinium Bromide | Placebo
Number analyzed (Participants) | 1791 | 1798
Participants
  Number of subjects with events | 69 | 76
Statistical Analysis 1: Comparison: Aclidinium Bromide vs Placebo; Composite MACE; Test type: Non-Inferiority — Estimate of the hazard ratio and its 95% CI for comparing aclidinium bromide 400 μg versus placebo were derived using the Cox proportional hazard model. A hazard ratio <1 represents a favorable outcome for aclidinium bromide 400 μg; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.64 to 1.23]

ADVERSE EVENTS:
Time Frame: Any adverse event occurring from the time the informed consent form was signed until 15 days after the last dose of study drug were recorded. Adverse events were collected at Visit 1A for subjects who completed a Visit 0.
Arm/Group | Aclidinium Bromide | Placebo
All-Cause Mortality (participants affected / at risk) | 75/1791 | 64/1798
Serious Adverse Events (participants affected / at risk) | 409/1791 | 356/1798
Other Adverse Events (participants affected / at risk) | 1105/1791 | 1065/1798
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide (N=1791) | Placebo (N=1798)
Appendicitis (Infections and infestations) | 5 (5) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 5 (6)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Infectious Colitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Breast Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Catheter Site Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 14 (16) | 10 (10)
Gangrene (Infections and infestations) | 0 (0) | 2 (2)
Meningitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 3 (3) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Breast Abscess (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter Colitis (Infections and infestations) | 0 (0) | 1 (1)
Extradural Abscess (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous Colitis (Infections and infestations) | 0 (0) | 1 (1)
Tongue Abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Lower Respiratory Tract Infection Fungal (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 0 (0) | 1 (1)
Post Procedural Infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Disease Carrier (Infections and infestations) | 0 (0) | 1 (1)
H1n1 Influenza (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 6 (6)
Pneumonia Influenzal (Infections and infestations) | 0 (0) | 1 (1)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 66 (78) | 58 (61)
Muscle Abscess (Infections and infestations) | 0 (0) | 1 (1)
Measles (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 12 (12) | 14 (14)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 5 (5) | 9 (10)
Gastroenteritis Viral (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0)
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Carcinoid Tumour Of The Stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dermatofibrosarcoma Protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of The Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Squamous Cell Carcinoma Of Head And Neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Lung Adenocarcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Adenocarcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6)
Non-Small Cell Lung Cancer Stage Iiib (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Respiratory Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Vaginal Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 3 (4)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (7)
Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Major Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 2 (2)
Alcohol Abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Drug Use Disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Substance Use Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Basal Ganglia Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 2 (2)
Cerebrovascular Accident (Nervous system disorders) | 9 (9) | 4 (4)
Embolic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 5 (5)
Lacunar Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Disease (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 4 (4) | 5 (6)
Balance Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 7 (7) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Tension Headache (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Hemianopia Homonymous (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 2 (4)
Radicular Pain (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Spinal Claudication (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 8 (9) | 5 (5)
Retinal Aneurysm (Eye disorders) | 1 (1) | 0 (0)
Retinal Artery Occlusion (Eye disorders) | 0 (0) | 2 (2)
Macular Fibrosis (Eye disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 2 (2) | 4 (5)
Atrioventricular Block Second Degree (Cardiac disorders) | 2 (2) | 0 (0)
Cardiovascular Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive Heart Disease (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 21 (22) | 8 (8)
Coronary Artery Occlusion (Cardiac disorders) | 2 (2) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac Failure Acute (Cardiac disorders) | 6 (6) | 6 (6)
Cardiac Failure Congestive (Cardiac disorders) | 21 (24) | 18 (19)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 14 (14) | 12 (12)
Angina Pectoris (Cardiac disorders) | 10 (10) | 9 (9)
Angina Unstable (Cardiac disorders) | 7 (7) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 10 (10) | 13 (13)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Bradycardia (Cardiac disorders) | 3 (3) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Right Ventricular Failure (Cardiac disorders) | 2 (2) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 24 (30) | 17 (22)
Atrial Flutter (Cardiac disorders) | 4 (4) | 3 (3)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Node Dysfunction (Cardiac disorders) | 0 (0) | 3 (3)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 3 (4)
Cardiac Arrest (Cardiac disorders) | 6 (6) | 4 (4)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Accelerated Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 2 (2)
Aortic Aneurysm (Vascular disorders) | 4 (4) | 2 (2)
Aortic Aneurysm Rupture (Vascular disorders) | 1 (1) | 1 (1)
Aortic Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Aortic Stenosis (Vascular disorders) | 2 (2) | 2 (2)
Leriche Syndrome (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic Shock (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Venous Disease (Vascular disorders) | 2 (2) | 0 (0)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 5 (5) | 2 (2)
Pelvic Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 3 (4) | 2 (2)
Intermittent Claudication (Vascular disorders) | 2 (2) | 1 (4)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 3 (5) | 3 (3)
Peripheral Artery Occlusion (Vascular disorders) | 0 (0) | 2 (2)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 1 (3)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Hypotension (Vascular disorders) | 8 (8) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 1 (1) | 0 (0)
Vena Cava Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 17 (18)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (13)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Thoracic Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 3 (4)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal Polyp Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis Ischaemic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 (5) | 4 (4)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 6 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's Oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal Food Impaction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 3 (3) | 3 (3)
Intestinal Ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestinal Stenosis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 (4) | 4 (4)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parotid Gland Enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis Acute (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 3 (3)
Jaundice Cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Bladder Diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder Necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 7 (7) | 7 (7)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal Failure (Renal and urinary disorders) | 5 (5) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Artery Thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Sudden Death (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 1 (1)
Systemic Inflammatory Response Syndrome (General disorders) | 2 (2) | 1 (1)
Mass (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 5 (5) | 3 (4)
Non-Cardiac Chest Pain (General disorders) | 17 (19) | 8 (10)
Electrocardiogram Abnormal (Investigations) | 0 (0) | 1 (1)
Heart Rate Decreased (Investigations) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 2 (2) | 2 (2)
Influenza A Virus Test Positive (Investigations) | 0 (0) | 1 (1)
Splenic Rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Coronary Vascular Graft Stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral Arterial Reocclusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Open Globe Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Femur Fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radial Head Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ulna Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve Root Injury Lumbar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Fat Embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Carbon Monoxide Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation Dysphagia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation Mucositis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured Sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Sternal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device Malfunction (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide (N=1791) | Placebo (N=1798)
Bronchitis (Infections and infestations) | 70 (85) | 74 (92)
Pneumonia (Infections and infestations) | 46 (51) | 52 (57)
Sinusitis (Infections and infestations) | 65 (87) | 63 (73)
Upper Respiratory Tract Infection (Infections and infestations) | 86 (104) | 101 (117)
Urinary Tract Infection (Infections and infestations) | 90 (122) | 84 (104)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 78 (95) | 67 (77)
Anaemia (Blood and lymphatic system disorders) | 40 (40) | 38 (39)
Headache (Nervous system disorders) | 57 (74) | 65 (84)
Dizziness (Nervous system disorders) | 44 (46) | 42 (45)
Atrial Fibrillation (Cardiac disorders) | 27 (30) | 40 (44)
Hypertension (Vascular disorders) | 64 (66) | 56 (60)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 (52) | 70 (74)
Cough (Respiratory, thoracic and mediastinal disorders) | 67 (71) | 62 (66)
Diarrhoea (Gastrointestinal disorders) | 58 (62) | 62 (67)
Constipation (Gastrointestinal disorders) | 60 (65) | 53 (53)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 38 (38) | 23 (23)
Nausea (Gastrointestinal disorders) | 77 (83) | 57 (64)
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 (53) | 45 (51)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 40 (44) | 34 (36)
Back Pain (Musculoskeletal and connective tissue disorders) | 69 (72) | 54 (57)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 28 (31) | 38 (40)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 35 (37) | 38 (41)
Oedema Peripheral (General disorders) | 48 (54) | 61 (70)
Anxiety (Psychiatric disorders) | 34 (35) | 39 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This submission /document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT01966107/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT01966107/SAP_001.pdf